CLINICAL TRIAL: NCT03509480
Title: Prospective Randomized Clinical Trial Comparing Ultraporous Beta-TCP With BMA to Combined TCP With Calcium Sulfate in Curetted Benign Bone Lesions
Brief Title: Vitoss With Bone Marrow Aspirate Versus Prodense
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Collaborators: Stryker Trauma and Extremities (Industry); Stryker Nordic (Industry)
Responsible Party: Principal Investigator, Timothy Damron, M.D., Professor, State University of New York - Upstate Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 248474
Record Dates: First submitted 2018-03-02; First posted 2018-04-26 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Bone Lesion

STUDY DESIGN:
Intervention Model Description: Comparison of ultraporous beta-tricalcium phosphate (Vitoss) with autologous bone marrow aspirate vs ultraporous beta-tricalcium phosphate with calcium sulfate (Prodense)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Curettage with Vitoss (Active Comparator): ultraporous beta-tricalcium phosphate mixed with autologous bone marrow aspirate for patients undergoing surgical curettage for benign bone lesions
  Interventions: Procedure: Surgical Curettage for benign bone lesion
- Curettage with Prodense (Active Comparator): ultraporous beta-tricalcium phosphate mixed with calcium sulfate for patients undergoing surgical curettage for benign bone lesions
  Interventions: Procedure: Surgical Curettage for benign bone lesion

INTERVENTIONS:
Procedure: Surgical Curettage for benign bone lesion — Surgical curettage for benign bone lesion, created defects will be filled with one of two types of graft material Vitoss versus Prodense, there are no other devices or drugs used

SUMMARY:
For benign curetted tumor defects, ultraporous beta-tricalcium phosphate (TCP) synthetic graft material (Vitoss; Orthovita, Inc., now Stryker, Inc.) persists for a year or longer in some cases even when BMA is added. What is not known is whether the addition to TCP of calcium sulfate (CS), which by itself has a more rapid resorption profile, will lead to more rapid resorption and incorporation of the composite graft material.

DETAILED DESCRIPTION:
Bone graft obtained from a patient's own bone (autogenous), usually around the pelvis, is currently considered the gold standard for bone grafting material. It provides a structural scaffold on which the patient's own bone may grow into (osteoconduction), growth factors that can stimulate healing (osteoinduction), and primitive cells (progenitors) that can stimulate bone formation directly (osteogenesis). It readily regains a blood supply from the surrounding tissues (revascularization) and is incorporated into the recipient site. However, there are significant disadvantages in the use of the patient's own bone graft including complications where the bone is taken from (donor site morbidity), limited availability and expense. Hence, human donor bone procured at the time of death (allografts) and synthetic bone fillers have been used as an alternative to the patient's own bone (autogenous bone graft). Both of these provide an osteoconductive scaffolding but nothing more. For defects created by scraping (curettage) of non-cancerous (benign) bone lesions, a structural scaffold (osteoconduction) is generally considered the minimal necessary role that the graft material must serve to allow healing of the defect. In many cases, this is adequate to allow healing of the defect by a process of creeping substitution, with neighboring bone growing from the periphery to the center in a centripetal fashion.

Ideally, the pace at which the graft material is resorbed is identical to the parallel pace of new bone formation. However, some materials have extremely slow replacement and are essentially never replaced fully for all practical purposes. An example of this is coralline hydroxyapatite. At the opposite end of the spectrum, some graft materials are resorbed at a far faster rate than bone formation. An example of this has been calcium sulfate. In the investigator's experience with the use of the synthetic bone graft substitute ultraporous beta-tricalcium phosphate (TCP) (Vitoss, Orthovita, Inc.) over the first 3 years of its availability, the graft material, when combined with local blood alone, performed well clinically but persisted for a year or longer radiographically in some cases. Prolonged persistence of the graft material may serve as a potential stress riser, although the investigator did not observe any untoward late effects in our published work. Subsequently, the investigator completed a randomized prospective evaluation of ultraporous beta-TCP alone and compared to beta-TCP combined with autologous bone marrow aspirate (BMA). The hypothesis was that both graft resorption and trabeculation (radiographic measures of incorporation of the synthetic material by the native bone) would be more advanced at each time point in those patients that received BMA plus TCP compared to those that received TCP alone. However, based upon the investigator's clinical impression, there does not appear to be a clinically relevant difference in the rate of bone incorporation. On the other hand, even at 1 year post-operatively, there appears by CT scan to be persistent beta-TCP in the grafted defects. Hence, it is felt that the rate of resorption and incorporation of the beta-TCP, with or without BMA does not keep pace with new bone formation.

Recently, a new osteoconductive synthetic bone graft material has become available that combines beta-TCP and calcium sulfate (PRO-DENSE® Injectable Regenerative Graft, Wright Medical Technology, Inc.). Theoretically, the calcium sulfate from this product will leach out more quickly, leaving a more porous local environment comprised of residual beta-TCP. Hence, the hypothesis of this study is that PRO-DENSE® may result in a more desirable, physiologic pace of graft incorporation when compared to beta-TCP and BMA. The overall study plan is to compare, in a randomized prospective fashion, PRO-DENSE injectable regenerative graft to ultraporous beta-TCP (VITOSS® morsels, OrthoVita, Inc.), the latter combined with bone marrow aspirate (BMA). VITOSS is the same porous material the investigator has used in an earlier study and is conducive to the addition of osteoinductive agents such as BMA, whereas PRO-DENSE is not.

A total of 56 patients with any type of benign bone lesion indicated for surgical curettage would be offered inclusion in the study, randomized to receive either PRO-DENSE or VITOSS with BMA, and followed for a minimum of 2 years post-operatively. Bone marrow aspiration would be obtained by a needle inserted through the skin (percutaneous aspiration) from the large bone of the pelvis (iliac crest) using a standard bone marrow aspiration needle. Patients with infection, bone marrow disorders, or other conditions that preclude use of supplementary the patient's bone marrow as well as those who prefer to use their own bone graft material (autograft) or donated human bone graft (allograft) alone would be excluded. Each patient will undergo radiographic evaluation of the lesion at 6 weeks, 3 months, 6 months, 1 year, 18 months and 2 years post operatively. At one time point (1 year) a computerized tomogram (CT) of the grafted region will be obtained for each patient. Two qualified, blinded, independent reviewers will evaluate the radiographs and CT scans for six criteria: 1.) presence of graft within the soft tissues, 2.) presence of a rim of radiolucency surrounding the grafted defect, 3.) size/circumference of the rim of radiolucency, 4.) resorption of graft material, 5.) trabeculation through the defect and 6.) persistence of graft material in the lesion. Kappa statistics have shown good agreement for these parameters in our published retrospective preliminary analysis of results for the TCP use without bone marrow by the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with cavitary bone lesions requiring surgical curettage (removal of tumor and scraping) will be asked to participate
* Patients must be able to read and understand the written informed consent
* Patients must be willing and able to return to the office for follow up appointments and xrays for at least two years

Exclusion Criteria:

* Patients with active or chronic infections
* Patients with bone marrow disorders
* Patients with contraindications to use of Vitoss or Prodense as listed on package inserts
* Patients who prefer to use autologous or allogeneic graft material alone (without synthetic filler)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Change in percentage of resorption of graft materials into the native bone as observed via CT scan | minimum of 24 months post operatively
  Radiographic interpretation by two independent radiologists was completed to assess the change in percentage of resorption of Vitoss with BMA or Prodense into the native bone at the 6 week, 3, 6, 12, 18 and 24 months timepoints based on review of x-ryas as well as by CT Scan at 12 month post operatively.

SECONDARY OUTCOMES:
Presence of graft material within the soft tissue | minimum of 24 months post operatively
  Radiographic interpretation by two independent radiologists was completed to assess presence of graft material within the soft tissue at the 6 week, 3, 6, 12, 18 and 24 months timepoints, based on radiograph and CT Scan review

OTHER OUTCOMES:
Change in presense (size/circumference) of radiolucency surrounding grafted defect | minimum of 24 months post operatively
  Radiographic interpretation by two independent radiologists was completed to assess change in presense (size/circumference) of radiolucency surrounding grafted defect at the 6 week, 3, 6, 12, 18 and 24 months timepoints, based on radiograph and CT Scan review
Change in trabeculation through the defect | minimum of 24 months post operatively
  Radiographic interpretation by two independent radiologists was completed to assess change in trabeculation (incorporation of graft into new bone) through the defect at the 6 week, 3, 6, 12, 18 and 24 months timepoints based on radiograph and CT Scan review
Change in persistence of graft material in the lesion | minimum of 24 months post operatively
  Radiographic interpretation by two independent radiologists was completed to assess the change in persistence of graft, how much graft material remains in the lesion at the 6 week, 3, 6, 12, 18 and 24 months timepoints based on radiograph and CT Scan review

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Damron, MD, Principal Investigator — SUNYUMU

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD at this time